CLINICAL TRIAL: NCT04441125
Title: The Effect of Labor Induction With Oxytocin on Early Postpartum Hemorrhage, Perineal Integrity and Breastfeeding
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Associate professor, Saglik Bilimleri Universitesi
Other Study IDs: 76
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Oxytocin
Keywords: Breastfeeding; Perineal Integrity; Postpartum Hemorrhage; oxytocin
MeSH Terms: conditions — Breast Feeding; Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: The mothers in the case group will receive oxytocin induction before and after delivery(n:44).
- control group: The mothers in the control group will not receive any oxytocin induction before delivery, and will receive oxytocin induction in the end of delivery(n:44)

SUMMARY:
Aim: This study has been planned as an observational study. The aim of this study is to determine the effect of labor induction with oxytocin on early postpartum hemorrhage, perineal integrity and breastfeeding.

Materials and Methods:

The sample consists of 88 healthy mother and infant pairs. The mothers in the case group will receive oxytocin induction before and after delivery. On the other hand, the mothers in the control group will not receive any oxytocin induction before delivery, and will receive oxytocin induction in the end of delivery.

Data were collected by using the Personal Information Form, the LATCH Breastfeeding Diagnostic Scale, the Breastfeeding Self-Efficacy Scale, the follow-up bag for postpartum hemorrhage, and episiotomy healing assessment known as the REEDA Scale.

DETAILED DESCRIPTION:
Oxytocin is applied to the women in the case group before the delivery.

There is a procedure on the usage of oxytocin at the delivery room. In accordance with the relevant procedure, it is administered as an intravenous infusion by adding 5 units of oxytocin in 500 cc of physiological saline solution.

The initial dosage is adjusted in order to allow for the flow of 4 drops per minute. Maximum 40 drops in total can be applied by increasing for 4 drops every 20 minutes. The dosage can be increased by considering the intensity and duration of contractions. The initial dosage of the oxytocin procedure applied to the women is the same for all women. As the total duration of delivery is different, there are differences between the dosages of oxytocin received.

In accordance with the postpartum procedure at the delivery room, it is administered as an intravenous infusion to all women (primiparous, multiparous) by adding 20 units of oxytocin in 500 cc of physiological saline solution immediately after the delivery.

The women in the control group do not receive any oxytocin induction before the delivery, and these women give birth spontaneously. After the delivery, the postpartum procedure applied for the control group is preferred.

Episiotomy is applied routinely to the primiparous pregnant women at the gynecological examination table in order to enlarge the opening of the vagina during the delivery. Episiotomy is a surgical incision applied to the bulbo-cavernous muscle in the perineal region while the baby's head appears in order to protect the perineal tonus, prevent undesired repairs, and to provide an easy, quick and safe delivery by enlarging the vaginal opening. Medio-lateral episiotomy is applied routinely to all women.

Immediately after the delivery, the baby's umbilical cord is clamped and cut. The postpartum hemorrhage bag is placed under the mother's perineal region immediately after the umbilical cord is cut, and it is waited for separation of the placenta. The duration for separation of the placenta is 30 minutes in maximum. After separation of the placenta, episiotomy repair is made. The loss of blood in the postpartum hemorrhage bag is recorded after the episiotomy repair. Before the woman is taken to her bed, necessary pads are provided, postpartum hemorrhage is followed-up, and the pads are weighed in the 24th postpartum hour.

The perineal region is evaluated by the REEDA scale in the postpartum 12th hour and the

The LATCH, the Breastfeeding Assessment, and the BSES are applied in the postpartum 24th hour and the first week.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 years,
* having a single pregnancy,
* literate,
* between 37-42 gestational week,
* hemoglobin level of 10 g and above,
* without chronic, mental and psychological disease

Infants;

* without congenital anomalies,
* with a first Apgar score of 8 and above,
* birth weight between 2500 - 4000 g
* no obstruction to oral feeding

Exclusion Criteria:

* multiparity,
* any risky condition development in the mother and baby during or after birth

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Women aged 18-35 years, having a single pregnancy, literate, between 37-42 gestational week, hemoglobin level of 10 g and above, without chronic, mental and psychological disease were included in the study. Infants without congenital anomalies, with a first Apgar score of 8 and above, birth weight between 2500- 4000 g and no obstruction to oral feeding constituted the sample of the study.
Study Population: The study consists of the primiparous pregnant women who comply with the study criteria, accept the study, and who are hospitalized in the delivery unit at Zeynep Kamil Women and Children Diseases Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
The REEDA (Redness, Oedema, Ecchymosis, Discharge and Approximation) | 12th hour
  Assessment is made by giving 0, 1, 2 and 3 scores to each title in the scale, and 0 is the lowest score and 15 is the highest score. 0 is the normal value for total score. In the scale, an increase in score indicates that there is pathology, and a decrease in score indicates that there is a recovery.
  The REEDA score is evaluated in the 12th hour after delivery.
The Breastfeeding Self-Efficacy Scale(BSES) | 24th hour
  This form is a five-point Likert-type scale, and it is scored as follows: "1=not at all confident", "2=not very confident", "3=sometimes confident", "4=confidentˮ, "5=very confidentˮ.
  The Breastfeeding Self-Efficacy Scale consists of 14 items.
  The lowest score which can be achieved from the scale is 14, and the highest score is 70.
  Achieving a high score indicates that the mothers have a high breastfeeding self-efficacy.
  The Breastfeeding Self-Efficacy is evaluated in the 24th hour after delivery.
L (LATCH on breast) A (Audible Swallowing) T (Type of Nipple) C (Comfort of Breast/Nipple) H (Hold/Positioni | 24th hour
  The LATCH: It consists of five evaluation criteria.
  Each item is evaluated between the score range of "0 - 2ˮ. In the scale, the highest score which can be achieved is 10, and the lowest score is 0. As the score achieved from this scale increases, the success in breastfeeding increases.
  The LATCH score is evaluated in the 24th hour after delivery.
The Follow-up Bag for Postpartum Hemorrhage(postpartum blood bag +pad weigth ) | 24th hour
  The postpartum hemorrhage bag has been calibrated in order to help for the follow-up of vaginal hemorrhage and fluid, and has been designed as filtration-specific. The bag is transparent colored, and the amount within the bag is recorded as milliliter.The postpartum hemorrhage bag is placed under the mother's perineal region after the delivery in order to measure the postpartum hemorrhage, and the amount of hemorrhage is recorded when the mother leaves the gynecological table. Then, the hemorrhage follow-up is made through a pad when the mother is taken to the bed. All pads are sterile and same in size. In the 24th postpartum hour, the pads used by the researcher are weighed and recorded.

SECONDARY OUTCOMES:
The REEDA (Redness, Oedema, Ecchymosis, Discharge and Approximation) | 24th hour
  Assessment is made by giving 0, 1, 2 and 3 scores to each title in the scale, and 0 is the lowest score and 15 is the highest score. 0 is the normal value for total score. In the scale, an increase in score indicates that there is pathology, and a decrease in score indicates that there is a recovery.
  The REEDA score is evaluated in the 24th hour after delivery.
The Breastfeeding Self-Efficacy Scale(BSES) | The first week
  This form is a five-point Likert-type scale, and it is scored as follows: "1=not at all confident", "2=not very confident", "3=sometimes confident", "4=confidentˮ, "5=very confidentˮ.
  The Breastfeeding Self-Efficacy Scale consists of 14 items.
  The lowest score which can be achieved from the scale is 14, and the highest score is 70.
  Achieving a high score indicates that the mothers have a high breastfeeding self-efficacy.
  The Breastfeeding Self-Efficacy is evaluated in the first week after delivery.
L (LATCH on breast) A (Audible Swallowing) T (Type of Nipple) C (Comfort of Breast/Nipple) H (Hold/Positioni | The first week
  The LATCH: It consists of five evaluation criteria.
  Each item is evaluated between the score range of "0 - 2ˮ. In the scale, the highest score which can be achieved is 10, and the lowest score is 0. As the score achieved from this scale increases, the success in breastfeeding increases.
  The LATCH score is evaluated in the first week after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: YASEMİN AYDIN KARTAL, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Zeynep Kamil Women's and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kartal YA, Kaya L, Yazici S. Effects of oxytocin induction on early postpartum hemorrhage, perineal integrity, and breastfeeding: a case-control study. Rev Assoc Med Bras (1992). 2023 Dec 22;70(1):e20231002. doi: 10.1590/1806-9282.20231002. eCollection 2023. PMID 38126414